CLINICAL TRIAL: NCT02224859
Title: Clinical Safety and Utility of the Invictus Cranial Support Device (CSD)
Brief Title: Invictus Medical, Medical Cranial Support Device (CSD) is a Device Safety Study in Infants at Risk of Head Ulcers.
Acronym: INV-CS-001
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Organization has withdrawn their 510k submission and stopped the study
Sponsor: Invictus Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: INV-CS-001; IND/IDE Number - IRB 013-306 (Other: Investigational Review Board - Baylor Health Care System)
Record Dates: First submitted 2014-03-28; First posted 2014-08-25 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Other Preterm Infants

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Safety (Other): Following an initial examination of the scalp and head for baseline evidence of skin integrity (intact, without breaks, lacerations, etc.) and appearance (healthy/normal, no erythema/irritation, etc.) the HCP will place the CSD on the patient and secure the attached Velcro strap to hold the device in place
  At specific time points (approximately 15 minutes, 1 hour, 3 hours and 6 hours) the HCP (through human intervention)will remove the CSD for examination and completion of the Skin Assessment Scale based on the appearance of the patient's scalp and adjacent areas of the head. Additionally, the patient's head will be observed for excessive scalp sweating/moisture accumulation.
  Interventions: Device: HCP will place the Invictus Cranial Support Device (CSD) on the patient; Other: human intervention

INTERVENTIONS:
Device: HCP will place the Invictus Cranial Support Device (CSD) on the patient — There is no active therapeutic treatment (e.g., medication, stimulation, etc.) associated with this device or study. All supplies for this study will be supplied by the sponsor and returned to them upon completion of the trial.
  The device used in this study is a soft gel based bonnet referred to as a Cranial Support Device (CSD). In this study, after obtaining written informed consent from the patient's parent(s) or guardian(s) and confirming that the patient meets all inclusion and no exclusion criteria, the study HCP will place the CSD on the selected patient.
Other: human intervention — This study is designed to evaluate the safety of the Invictus Cranial Support Device (CSD) when worn by medically stable infants within a neonatal intensive care unit (NICU), to evaluate the form, fit, and ease of use/application of the CSD device (i.e., utility), as well as initial impressions of safety, by health care providers (HCPs) after placing the current CSD on infants for approximately six (6) hours in a NICU

SUMMARY:
While using the device as a cushion, the passive distribution of pressure over bony skull prominences of infants will protect against formation of pressure ulcers.

DETAILED DESCRIPTION:
This study is designed to evaluate the safety of the Invictus Cranial Support Device (CSD) when worn by medically stable infants within a neonatal intensive care unit (NICU), to evaluate the form, fit, and ease of use/application of the CSD device (i.e., utility), as well as initial impressions of safety, by health care providers (HCPs) after placing the current CSD on infants for approximately six (6) hours in a NICU. Specifically, this study will:

* Collect safety information at specified time points (baseline, 15 minutes, 1 hour, 3 hours, and 6 hours) utilizing a widely used dermal assessment tool, health assessments (temperature, pulse, respiration rate), excessive scalp sweating/moisture accumulation, and adverse events, as reflected in the Table 1.0, Time and Events Table.

Additional safety assessments will be performed following the final removal of the CSD from the infants head. Refer to Table 1.0 Time and Events Table and section 6.1.

* Assess the HCP's impression of likely safety and effectiveness (Function Assessments) of the CSD based on experience working with infants in the NICU, Evaluate/Rate the form and fit, and evaluate/rate the ease of application of the product.
* Collect additional feedback (if any) on HCP's impressions of device design and usability based on experience working as a HCP in the NICU

ELIGIBILITY:
Inclusion Criteria:

1. Have a parent(s) or guardian(s) who has provided written informed consent for the patient to participate in the study.
2. Be > 30.0 weeks gestational age at time of enrollment into the study
3. Be in medically stable condition within the NICU
4. Be able to breathe adequately on room air without support
5. Be deemed suitable (i.e., in no acute distress) for participating in the study for approximately six (6) hours, in the investigator's opinion
6. Upon visual inspection have intact skin without breaks and/or lacerations of the scalp or adjacent areas where the CSD will fit

Exclusion Criteria:

1. The use of any additional respiratory support (i.e., intubation, using CPAP, etc.) is required,
2. The patient has any genetic dermatological conditions
3. The patient's head size is not appropriate for the device < 28 centimeters or >34.3 centimeters (< 11 or > 13.5 inches)
4. Patient has significant medical condition(s) (e.g., encephalocele, IVH, Shunt, etc.) that makes participating in the study not in the patient's best interest

Ages: 30 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2014-03; Primary Completion 2015-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
HCP assessments of the products form, fit, likely effectiveness, and safety for internal decision making and for support of an FDA 510K submission to demonstrate form and fit as it relates to a predicate device. | Each patient will spend approximately six (6) hours in the study if no adverse experiences
  Rating scale data will be collected and analyzed using descriptive statistics to determine overall HCP assessments of the products form, fit, likely effectiveness, and safety for internal decision making and for support of an FDA 510K submission to demonstrate form and fit as it relates to a predicate device. No hypothesis testing will be conducted. Only descriptive statistics, frequency counts, and proportions will be used to summarize the data. Descriptive statistics, such as number of observations, means, standard deviations, medians, and maximum and minimum values, will be used to summarize the continuous variables. Frequencies and proportions will be used to summarize categorical variables.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa . Suterwala, MD, Principal Investigator — Baylor Health Care System
Locations (1):
- Baylor University Medical Center, Dallas, Texas, United States